CLINICAL TRIAL: NCT05564312
Title: The Effect of Embryo Transfer Technique on Pregnancy Outcomes in HRT-FET Cycles Using High-Quality Blastocyst Stage Embryos: a Prospective Cohort Study
Brief Title: The Effect of Embryo Transfer Technique on Pregnancy Outcomes in HRT-FET Cycles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, Associate Professor, Akdeniz University
Other Study IDs: 49829699
Record Dates: First submitted 2022-09-29; First posted 2022-10-03 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Infertility
Keywords: air bubble position; embryo transfer; ultrasonographic guidance
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- non-pregnant: Negative b-hCG results 9 days after embryo transfer.
  Interventions: Device: Transabdominal ultrasonographic guidance at embryo transfer.
- pregnant: Positive b-hCG results 9 days after embryo transfer.
  Interventions: Device: Transabdominal ultrasonographic guidance at embryo transfer.

INTERVENTIONS:
Device: Transabdominal ultrasonographic guidance at embryo transfer. — During embryo transfer in each patient, endometrial thickness, uterine cavity dimensions, distance of transfer catheter to the fundus, distance of released air bubble to the fundus, and distance of air bubble to side walls will be systematically measured and recorded under the guidance of transabdominal ultrasonography.

SUMMARY:
The positions of the air bubble and the tip of catheter will be measured by transabdominal utrasonography among patients who have undergone high-quality frozen blastocyst transfer. The aim of this study is to compare pregnancy rates according to air bubble's final location in endometrial cavity. It is expected that the ET technique will be improved and live birth rates will increase by determining the optimal position of the embryo in the endometrial cavity during ET in patients who have achieved pregnancy.

DETAILED DESCRIPTION:
Only patients who have high-quality blastocyst stage embryos will be included in the study. Since the implantation potential of high-quality embryos is high, possible embryo-induced implantation failure will be minimized. The positions of the air bubble and the catheter in the endometrial cavity in patients with and without pregnancy will be compared.

In patients participating in the study, the transfer catheter will be loaded using a "three drop technique," in which the drop of medium containing the embryo(s) is/are separated from a preceding and a following drop of the medium by an air bubble.

In hormonally prepared frozen embryo cycles, during embryo transfer in each patient, endometrial thickness, uterine cavity dimensions, distance of transfer catheter to the fundus, distance of released air bubble to the fundus, and distance of air bubble to side walls will be systematically measured and recorded under the guidance of transabdominal ultrasonography.

If the position of the embryo in the endometrial cavity is determined during ET in patients who have achieved pregnancy, an ET technique can be defined that predicts the optimum for the physician who will perform the transfer. Therefore, an increase in implantation and pregnancy rates can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Exogenous hormone preparation of the endometrial lining
* High embryo quality ((≥2BB) according to Alpha criteria
* Embryo transfer at the blastocyst stage

Exclusion Criteria:

* Patients whose treatments were canceled for any reason before the embryo transfer procedure
* Patients who underwent embryo transfer in the cleavage stage
* Presence of low-quality (<2BB) blastocysts
* >15% loss of viability of the embryo during embryo thawing,
* Patients with congenital uterine malformations,

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: All patients who have artificial endometrial preparation with high-quality blastocysts between December 2021 and December 2022 will be included.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Positive β-hCG results | Nine days after each embryo transfer
  Positive β-hCG results nine days after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: ŞAFAK OLGAN, MD, Principal Investigator — Akdeniz University; ARİF C ÖZSİPAHİ, MD, Study Chair — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)